CLINICAL TRIAL: NCT01262053
Title: Investigating Wrong-Patient CPOE Errors
Brief Title: Investigating Wrong-Patient Computerized Physician Order Entry (CPOE) Errors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 10-05-156E
Record Dates: First submitted 2010-12-15; First posted 2010-12-17 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Wrong Patient Computerized Physician Order Entry Errors
Keywords: Computerized Physician Order Entry; CPOE; Wrong Patient; Juxtaposition; Patient Safety; Medical Errors

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Passive Intervention (Experimental): When a user is about to place orders on a patient, a pop up alert will show the user the name, age, sex, room number and MR# of the patient who is currently activated.
  Interventions: Other: Passive Intervention
- Active Intervention (Experimental): The user will be required to enter the initials, age and sex of the activated patient prior to placing any orders.
  Interventions: Other: Active Intervention
- Control (Active Comparator): Parallel control with no intervention
  Interventions: Other: Control

INTERVENTIONS:
Other: Passive Intervention — When a user is about to place orders on a patient, a pop up alert will show the user the name, age, sex, room number and MR# of the patient who is currently activated. The point of the alert is to display identification information about the patient as a double check for the provider to make sure he is on the correct patient. This alert will only occur once at the onset of each order session (i.e. the provider will not be alerted for every single order, but if the provider leaves the order pad and then returns, the alert will reoccur).
  Arms: Passive Intervention
Other: Active Intervention — The user will be required to enter the initials, age and sex of the activated patient prior to placing any orders. For example, for a patient named Donald Duck who is 76 years old and male, the user will be required to type "dd76m" to unlock the order pad. This step will NOT be required for every order, but WILL be required every time the user enters the order pad (i.e. if a user leaves the order pad and then returns, the system will require the initials, age and sex to be re-entered as above). This will be a forcing function.
  Arms: Active Intervention
Other: Control — Parallel control with no intervention
  Arms: Control

SUMMARY:
With the increased adoption of CPOE systems, it is important to recognize that design flaws have resulted in the creation of new types of iatrogenic medical errors. An example of a new type of iatrogenic medical error introduced by CPOE systems has been named "juxtaposition errors". Juxtaposition errors, as defined by Ash, et al. are "errors that can result when something is close to something else on the screen, and the wrong option is too easily clicked in error." Juxtaposition errors can lead to a patient receiving a medication, a test, or a treatment intended for another patient, sometimes with dire consequences. Juxtaposition errors are likely a subclass of a broader group of wrong-patient CPOE errors that have multiple etiologies.

The primary objectives of this research proposal is to investigate the prevalence of wrong-patient near miss CPOE errors, to investigate the root cause of these errors, and to investigate and compare the efficacy and workflow impact of two distinct interventions to prevent these errors.

DETAILED DESCRIPTION:
Computerized Physician Order Entry (CPOE) systems have been shown to prevent medical errors, and have become a major component of the patient safety movement. To accelerate the adoption of clinical information technology including CPOE systems, the American Recovery and Reinvestment Act of 2009 allocated approximately $17 billion as incentive payments to providers and hospitals who implement health information technology. With the increased adoption of CPOE systems, however, it is important to recognize that design flaws have resulted in the creation of new types of iatrogenic medical errors. In addition, CPOE systems developed with suboptimal and onerous user interfaces have contributed to entire systems being rejected by physicians. The ideal CPOE system maximizes medical error reduction, minimizes medical error creation, and has a user friendly interface that is accepted by nurses, physicians, and pharmacists.

An example of a new type of iatrogenic medical error introduced by CPOE systems has been named "juxtaposition errors" . Juxtaposition errors, as defined by Ash, et al. are "errors that can result when something is close to something else on the screen, and the wrong option is too easily clicked in error." Juxtaposition errors can lead to a patient receiving a medication, a test, or a treatment intended for another patient, sometimes with dire consequences.

Juxtaposition errors are likely a subclass of a broader group of wrong-patient CPOE errors that have multiple etiologies. Other possible causes of wrong-patient CPOE orders include interruption errors, or double-interruption errors.

Primary Objectives:

* Specific Aim 1: Investigate the prevalence of wrong-patient near miss CPOE errors.
* Specific Aim 2: Investigate the root cause of wrong-patient near miss CPOE errors.
* Specific Aim 3: Investigate and compare the efficacy and workflow impact of two distinct interventions to prevent wrong-patient near miss CPOE errors against a control.

ELIGIBILITY:
Inclusion Criteria:

* All providers that place order in the Computerized Physician Order Entry (CPOE) System

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4028 (Actual)
Dates: Start 2010-12; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Reduction of wrong patient CPOE errors | Within one hour of placing an order
  Compare reduction of wrong patient CPOE errors in each intervention group against a control

SECONDARY OUTCOMES:
Impact of interventions on workflow | Within one hour of placing an order
  Compare the efficacy and workflow impact of two distinct interventions to prevent wrong-patient near miss CPOE errors against a control

CONTACTS AND LOCATIONS:
Overall Officials: Jason S Adelman, MD, MS, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ash JS, Sittig DF, Poon EG, Guappone K, Campbell E, Dykstra RH. The extent and importance of unintended consequences related to computerized provider order entry. J Am Med Inform Assoc. 2007 Jul-Aug;14(4):415-23. doi: 10.1197/jamia.M2373. Epub 2007 Apr 25. PMID 17460127
- [Background] Koppel R, Metlay JP, Cohen A, Abaluck B, Localio AR, Kimmel SE, Strom BL. Role of computerized physician order entry systems in facilitating medication errors. JAMA. 2005 Mar 9;293(10):1197-203. doi: 10.1001/jama.293.10.1197. PMID 15755942
- [Background] Weiner JP, Kfuri T, Chan K, Fowles JB. "e-Iatrogenesis": the most critical unintended consequence of CPOE and other HIT. J Am Med Inform Assoc. 2007 May-Jun;14(3):387-8; discussion 389. doi: 10.1197/jamia.M2338. Epub 2007 Feb 28. No abstract available. PMID 17329719
- [Background] Campbell EM, Sittig DF, Ash JS, Guappone KP, Dykstra RH. Types of unintended consequences related to computerized provider order entry. J Am Med Inform Assoc. 2006 Sep-Oct;13(5):547-56. doi: 10.1197/jamia.M2042. Epub 2006 Jun 23. PMID 16799128
- [Background] Wachter RM. Expected and unanticipated consequences of the quality and information technology revolutions. JAMA. 2006 Jun 21;295(23):2780-3. doi: 10.1001/jama.295.23.2780. No abstract available. PMID 16788133